CLINICAL TRIAL: NCT00077766
Title: A Randomized, Controlled, Open-label, Multi-center, Parallel-group Study to Demonstrate the Efficacy and Safety of RO0503821 When Administered Intravenously for the Maintenance Treatment of Anemia in Patients With Chronic Kidney Disease Who Are on Dialysis.
Brief Title: A Study of Intravenous Mircera for the Treatment of Anemia in Dialysis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA17283
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Results first posted 2016-09-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2015-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; continuous erythropoietin receptor activator

ARMS (2):
- RO0503821 (1x/2 Weeks) (Experimental): Eligible participants will be administered with RO0503821 ([methoxy polyethylene glycol-epoetin beta] {Mircera}) intravenously (IV), every 2 weeks during Weeks 1 through 52. The starting dose of RO0503821 (60, 100, or 180 micro gram [µg]) was based on the dose of darbepoetin alfa at the time of randomization (< 40, 40 to 80, or > 80 µg per week, respectively).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Darbepoetin (1x/1-2 Weeks) (Active Comparator): Eligible participants will be administered with darbepoetin alfa IV, every week or every 2 weeks during Weeks 1 through 52.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoetin alfa was administered IV, every week or every 2 weeks during Weeks 1 through 52.
  Arms: Darbepoetin (1x/1-2 Weeks)
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — RO0503821 was administered IV, every 2 weeks during Weeks 1 through 52. The starting dose of RO0503821 (60, 100, or 180 micro gram [µg]) was based on the dose of darbepoetin alfa at the time of randomization (< 40, 40 to 80, or > 80 µg per week, respectively).
  Arms: RO0503821 (1x/2 Weeks)

SUMMARY:
This study will assess the efficacy and safety of intravenous (iv) Mircera given as maintenance treatment for renal anemia in chronic kidney disease patients on dialysis who were previously receiving iv darbepoetin alfa. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* on dialysis therapy for at least 12 weeks before screening;
* receiving darbepoetin alfa iv for at least 8 weeks before screening.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of another investigational drug within 4 weeks before screening, or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2004-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (47):
- Australia (6):
  - Blacktown
  - Brisbane
  - Clayton
  - Gosford
  - Parkville
  - Sydney
- Graz, Austria
- Belgium (3):
  - Aalst
  - Brussels
  - Liège
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kamloops, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Kitchener, Ontario
  - Mississauga, Ontario
- Denmark (3):
  - Aalborg
  - Odense
  - Roskilde
- HUS, Finland
- France (6):
  - Aubervilliers
  - Montpellier
  - Nice
  - Strasbourg
  - Tarbes
  - Toulouse
- Germany (3):
  - Hannoversch Münden
  - Nuremberg
  - Villingen-Schwenningen
- Italy (5):
  - Bergamo
  - Lecco
  - Livorno
  - Messina
  - Pavia
- Spain (7):
  - Badalona
  - Barcelona
  - Córdoba
  - Madrid
  - Oviedo
  - Salamanca
  - Santander
- Sweden (2):
  - Karlstad
  - Stockholm
- Switzerland (2):
  - Aarau
  - Lausanne

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Canaud B, Mingardi G, Braun J, Aljama P, Kerr PG, Locatelli F, Villa G, Van Vlem B, McMahon AW, Kerloeguen C, Beyer U; STRIATA Study Investigators. Intravenous C.E.R.A. maintains stable haemoglobin levels in patients on dialysis previously treated with darbepoetin alfa: results from STRIATA, a randomized phase III study. Nephrol Dial Transplant. 2008 Nov;23(11):3654-61. doi: 10.1093/ndt/gfn320. Epub 2008 Jun 27. PMID 18586762

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 313 participants were randomized in this study conducted from 10 March 2004 to 31 August 2005 in 12 countries.
Groups:
- RO0503821 (1x/2 Weeks): Eligible participants were administered with RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) intravenously (IV), every 2 weeks during Week 1 through Week 52. The starting dose of RO0503821 (60, 100, or 180 microgram [µg]) was based on the dose of darbepoetin alfa at the time of randomization (< 40, 40 to 80, or > 80 µg per week, respectively).
- Darbepoetin (1x/1-2 Weeks): Eligible participants were administered with darbepoetin alfa IV, every week or every 2 weeks during Week 1 through Week 52.
Period: Overall Study
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Started | 157 | 156
Completed | 118 | 131
Not Completed | 39 | 25
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 12 | 10
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Kidney Transplantation | 9 | 5
Not completed — Transplantation | 5 | 1
Not completed — Investigators Discretion | 1 | 0
Not completed — Participant's decision | 1 | 0
Not completed — Dialysis Discontinued | 1 | 0
Not completed — Dialysis | 0 | 1
Not completed — Enrolled in Nocturnal Hemodialysis Study | 0 | 1
Not completed — Started Nocturnal Dialysis | 0 | 1
Not completed — Stop Dialysis | 0 | 1
Not completed — Participants Vacation | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants who received at least one dose of RO0503821 or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. There were 4 participants who were excluded from the safety population as they did not receive the study medication.
Groups:
- RO0503821 (1x/2 Weeks): Eligible participants were administered with RO0503821 IV, every 2 weeks during Week 1 through Week 52. The starting dose of RO0503821 (60, 100, or 180 µg) was based on the dose of darbepoetin alfa at the time of randomization (< 40, 40 to 80, or > 80 µg per week, respectively).
- Total: Total of all reporting groups
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks) | Total
Number analyzed (Participants) | 153 | 156 | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (15.72) | 61.9 (14.74) | 62.2 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 74 | 130
  Male | 97 | 82 | 179

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Concentration (g/dL) From Baseline to Evaluation Period
Description: A time adjusted mean change in hemoglobin (Hb) concentration was calculated using an area under the curve approach, for both periods separately. Change in Hb concentration between the baseline (Week -4 to Week -1) and evaluation periods was calculated by subtracting the calculated average baseline Hb value from the average evaluation period Hb value. All blood samples for Hb measurements were taken prior to study drug administration. The analysis used the last observation carried forward (LOCF) for missing Hb values for correction of the impact of early drop outs. The baseline period was defined as Week -4 to Week -1. The evaluation period was defined as Week 29 to Week 36.
Time Frame: Baseline (Week -4 to Week -1) and Evaluation Period (Week 29 to Week 36)
Population: The per protocol population was all randomized and treated participants, except those who had not met criteria for stable baseline Hb,and adequate iron levels or had hemoglobinopathies/hemolysis, RBC transfusion/blood loss, <5 recorded Hb values during evaluation or missed administrations of trial drugs in week 26 to 35.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Groups:
- RO0503821 (1x/2 Weeks): Eligible participants were administered with RO0503821 IV, every 2 weeks during Weeks 1 through 52. The starting dose of RO0503821 (60, 100, or 180 µg) was based on the dose of darbepoetin alfa at the time of randomization (< 40, 40 to 80, or > 80 µg per week, respectively).
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 123 | 126
gram per deciliter (g/dL) | 0.05 (0.96) | -0.10 (0.92)
Statistical Analysis 1: Comparison: RO0503821 (1x/2 Weeks) vs Darbepoetin (1x/1-2 Weeks); RO0503821 group was compared to darbepoetin alfa group, using analysis of covariance (ANCOVA) with the independent variable as treatment group and Hb at baseline and geographical region as covariates. The test for non-inferiority was based on the lower limit of 2-sided 95% confidence interval (CI) for difference in adjusted mean between 2 groups. If this lower limit was > or = to -0.75 g/dL, the RO0503821 group was regarded as clinically non-inferior to darbepoetin alfa group, with 90% power; Test type: Non-Inferiority or Equivalence — Non-inferiority with 90% power assuming that the true difference between the RO0503821 group and darbepoetin was not larger than 0.3 g/dL; p < 0.0001, ANCOVA, CI for difference between groups — The p-value for the non-inferiority test was derived using ANCOVA; Degrees of Freedom : 246; Mean Difference (Final Values) = 0.180, 95% CI 2-sided [-0.049 to 0.408], Standard Error of Mean 0.1162 — Difference between groups based on the adjusted means derived from the ANCOVA model

2. Secondary Outcome: Number of Participants Maintaining Average Hemoglobin Concentration During the Evaluation Period Within +-1 g/dL of Their Average Baseline Hemoglobin Concentration
Description: The average Hb of all values recorded during the evaluation period was calculated, and this average was subtracted from the average baseline Hb values for each participant. The number of participants maintaining their average Hb within +/- 1 g/dL of their average baseline Hb concentration is displayed. The evaluation period was defined as Week 29 to Week 36.
Time Frame: Baseline (Week -4 to Week -1) and Evaluation Period (Week 29 to Week 36)
Population: The Intent-to-Treat (ITT) population was defined as all randomized participants. Participants with available data at the time of evaluation were analyzed.
Measure: Number; unit: Participants
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 139 | 142
Participants | 91 | 102

3. Secondary Outcome: Number of Participants With Red Blood Cell Transfusions During the Dose Titration and Evaluation Periods
Description: A combined data of the number of participants who received Red Blood Cell (RBC) transfusions during the titration and evaluation periods is reported. A period of 28 weeks after the first dose of the study drug was used for dose titration and stabilization of Hb concentration. The dose titration period was followed by an 8-week evaluation period (weeks 29 to 36).
Time Frame: Week 1 to Week 36
Population: The safety population was defined as all participants who received at least one dose of RO0503821 or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not.
Measure: Number; unit: Participants
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 153 | 156
Participants | 19 | 16

4. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: A marked abnormality range was defined as above and/or below a value which was considered to be potentially clinically relevant. Marked laboratory abnormalities were analyzed according to the Roche specified limits for the reference range of the following laboratory parameters: White blood cells (WBC) (3.0- 18.0 10^9/liter [L]), platelets (100 - 550 10^9/L), (alanine aminotransferase [(ALAT)] (0 - 110 units per liter [U/L]), alkaline phosphatase (ALP) (0 - 220 U/L), aspartate aminotransferase (ASAT) (0 - 80 U/L), albumin >= 30 g/L, phosphate (0.75 - 1.60 millimole per liter [mmol/L]), potassium (2.9 - 5.8 mmol/L), glucose (2.80 - 11.10 mmol/L).
Time Frame: Up to Week 52
Population: The safety population was defined as all participants who received at least one dose of RO0503821 or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. Data from participants available at protocol specified assessment time points were included in the analysis (n).
Measure: Number; unit: Participants
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 152 | 154
Participants
  Platelets, High; n=152,153 | 0 | 6
  Platelets, Low; n=152,153 | 6 | 4
  WBC, High; n=152,153 | 4 | 3
  WBC, Low; n=152,153 | 6 | 4
  ALAT, high; n=152,154 | 4 | 2
  ALP, High; n=152,154 | 6 | 11
  ASAT, High; n=148,151 | 7 | 5
  Albumin, Low; n=143,142 | 12 | 14
  Phosphate, High; n=152,154 | 60 | 61
  Phosphate, Low; n=152,154 | 9 | 13
  Potassium, High; n=152,154 | 38 | 31
  Potassium, Low; n=152,154 | 0 | 1
  Glucose (fasting), High; n=103,100 | 1 | 0

5. Secondary Outcome: Mean Change in Blood Pressure From Baseline at Week 36 and Week 52
Description: Blood pressure Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) was measured by manual assessment or automated reading throughout the study for every participant. Blood pressure was taken in the sitting position after at least 5 minutes rest. An appropriate -sized cuff was used and both systolic and diastolic blood pressures were recorded before dialysis (BD) and after dialysis (AD).
Time Frame: Baseline, Week 36, and Week 52
Population: The safety population was defined as all participants who received at least one dose of RO0503821 or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. Data from participants available at protocol specified assessment time point were included in the analysis (n).
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 130 | 134
millimeters of mercury (mm Hg)
  Change in SBP, BD, at Week 36, n = 130, 134 | -2 (23.0) | -2 (24.3)
  Change in DBP, BD, at Week 36, n = 130, 134 | -0 (12.8) | -2 (16.4)
  Change in SBP, BD, at Week 52, n = 117, 130 | 2 (24.6) | -4 (22.0)
  Change in DBP, BD, at Week 52, n = 117,130 | 0 (12.4) | -3 (16.0)
  Change in SBP, AD, at Week 36, n = 130, 132 | -3 (25.9) | -3 (24.0)
  Change in DBP, AD, at Week 36, n = 130, 132 | -3 (13.6) | -4 (14.2)
  Change in SBP, AD, at Week 52, n = 116,129 | -0 (26.9) | -3 (25.0)
  Change in DBP, AD, at Week 52, n = 116,129 | -1 (15.0) | -4 (14.9)

6. Secondary Outcome: Mean Change in Pulse Rate (Sitting) From Baseline at Week 36 and Week 52
Description: Change in pulse rate (beats per minute [bpm]) from baseline values includes only those participants with both a baseline (BL) value and a value for specified time period.
Time Frame: Baseline, Week 36, and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 126 | 128
beats per minute
  Change From Baseline to Week 36, n=126, 128 | -1 (11.9) | 1 (10.6)
  Change From Baseline to Week 52, n=112, 126 | -1 (13.0) | 0 (13.5)

7. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Event, and Deaths
Description: An Adverse Event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes. Overall deaths occurred in the study were reported.
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Number analyzed (Participants) | 153 | 156
Participants
  Number of participants with any AEs | 135 | 143
  Number of participants with any SAEs | 71 | 75
  Number of deaths (all causes) | 13 | 12

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: AE is untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event is with any of the following outcomes: Death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity; congenital anomaly.
Arm/Group | RO0503821 (1x/2 Weeks) | Darbepoetin (1x/1-2 Weeks)
Serious Adverse Events (participants affected / at risk) | 71/153 | 75/156
Other Adverse Events (participants affected / at risk) | 97/153 | 93/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/2 Weeks) (N=153) | Darbepoetin (1x/1-2 Weeks) (N=156)
Pneumonia (Infections and infestations) | 7 | 7
Sepsis (Infections and infestations) | 2 | 3
Bacteraemia (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 2 | 1
Arteriovenous graft site Infection (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 0 | 2
Infected skin ulcer (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Lower respiratory tract (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 1
Staphylococal infection (Infections and infestations) | 0 | 2
Bronchitis acute (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter sepsis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 0 | 1
Diabetic Gangrene (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Injection site infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Localized infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Postoperative infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 1
Arteriovenous fistula (Injury, poisoning and procedural complications) | 5 | 4
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 | 5
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Treatment compliance (Injury, poisoning and procedural complications) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 2
Angina pectoris (Cardiac disorders) | 3 | 2
Cardiac arrest (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Cardiac disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dizzinesss (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoasthesia (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 2 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 3
Peripheral ischaemia (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arteriopathic disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 2
Chest pain (General disorders) | 2 | 0
Hyperpyrexia (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Catheter related complication (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Disability (Social circumstances) | 0 | 1
Corneal transplant (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/2 Weeks) (N=153) | Darbepoetin (1x/1-2 Weeks) (N=156)
Diarrhoea (Gastrointestinal disorders) | 23 | 15
Vomiting (Gastrointestinal disorders) | 10 | 13
Nausea (Gastrointestinal disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 9 | 4
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3
Nasopharyngitis (Infections and infestations) | 19 | 16
Influenza (Infections and infestations) | 19 | 11
Upper respiratory tract infection (Infections and infestations) | 9 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 8
Hypertension (Vascular disorders) | 12 | 12
Hypotension (Vascular disorders) | 8 | 5
Haematoma (Vascular disorders) | 2 | 8
Wound (Injury, poisoning and procedural complications) | 9 | 6
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 8 | 6
Procedural hypotension (Injury, poisoning and procedural complications) | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Fluid overload (Metabolism and nutrition disorders) | 12 | 11
Headache (Nervous system disorders) | 8 | 12
Pyrexia (General disorders) | 10 | 6
Angina pectoris (Cardiac disorders) | 9 | 6
Depression (Psychiatric disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.